CLINICAL TRIAL: NCT05057884
Title: Breathing Exercise Against Dyspnoea in Heart Failure Patients to Improve Chemosensitivity and Ventilatory Efficiency - a Randomized Controlled Single-centre Trial
Brief Title: Breathing Exercise Against Dyspnoea in Heart Failure Patients to Improve Chemosensitivity
Acronym: Breathe-HF
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of finances
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Breathe-HF
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing training (Experimental): The respiratory pattern modulation training is performed at home for 12 weeks twice daily for 15 min per session and consists of three components: 1) education on abnormal ventilation in heart failure, the effect of ventilation on PaCO2 and the autonomous nervous system, and chemoreceptor sensitivity; 2) 1-3 sessions of guided and monitored face-to-face training with slow nasal abdominal breathing and intermittent apnoea supported by the Healer vest (L.I.F.E., Milan, Italy) measuring electrocardiogram (ECG), and chest excursions at the level of the xiphoid, thoracic manubrium, and abdomen; 3) independent home-based apnoea training supported by hand-outs, videos and weekly phone calls to monitor progress and adherence, answer questions and encourage further progression with duration of breath-hold.
  Interventions: Behavioral: Breathing training
- Control (No Intervention): The control group receives standard of care. They perform the study measurements before and after the intervention period of 12 weeks. They are offered to perform the breathing training after study completion.

INTERVENTIONS:
Behavioral: Breathing training — Slow nasal breathing with intermittent end-expiratory apnoea for 15 min twice per day over 12 weeks.
  Arms: Breathing training

SUMMARY:
An exaggerated ventilatory response (minute ventilation, V̇E) to exercise relative to exhaled carbon dioxide (V̇CO2) is common in heart failure (HF) patients with reduced as well as preserved left ventricular ejection fraction (HFrEF, HFpEF). Severity of this exaggerated response is associated with poor prognosis. This response may be triggered by pulmonary congestion and peripheral muscle myopathy. A vicious circle is fuelled by hypersensitivity of chemoreceptors to hypercapnia and sympathetic nervous hyperactivity, resulting in hyperventilation (low PaCO2). Low PaCO2 is predictive of mortality in these patients. PaCO2 can be increased acutely, e.g. by apnoea. Also, nasal breathing has been found to reduce the V̇E/V̇CO2 slope during exercise compared to oral breathing. Three previous slow breathing studies in HFrEF patients have had encouraging results with regard to reducing sympathetic activity, reflected in lowered arterial (pulmonary) blood pressure and increased EF. The investigators hypothesise that a 12-week training with nasal slow breathing followed by end-expiratory apnoea based on education, centre-based introduction and home-based 15 min/day breathing training will be effective at reducing the exaggerated ventilatory response to exercise. A total of 68 patients with stable HF seen at the HF clinics of the Inselspital (34 HFrEF, 34 HFpEF) will be randomised to the breathing intervention or usual care. Primary outcome will be V̇E/V̇CO2 slope at 12 weeks. If breathing training successfully ameliorates the exaggerated ventilatory response and perception of dyspnea during exercise, it offers an attractive tele-health based add-on therapy that may add to or even amplify the beneficial effects of exercise training.

DETAILED DESCRIPTION:
BACKGROUND

Ventilatory inefficiency, most commonly quantified as an increased ventilation (V̇E) to carbon dioxide exhalation (V̇CO2) slope during exercise, is a landmark of heart failure patients both with reduced and preserved ejection fraction (HFrEF, HFpEF).[1] Numerous studies have found higher V̇E/V̇CO2 slopes to be associated with poorer prognosis.[2-4] The components of the V̇E/V̇CO2 slope are the arterial CO2 partial pressure (PaCO2), that is affected by hyperventilation, and the pulmonary dead space/tidal volume ratio (VD/VT) that is affected by pulmonary perfusion abnormalities.[5] The exaggerated response in ventilation of HFrEF patients may be caused by hypersensitivity of chemoreceptors to CO2,[6] and/or a sympathetic nervous hyperactivity commonly found in HFrEF patients, based on an increased activation of metaboreceptors in peripheral muscles response to increased anaerobic metabolism.[7] Chronic sympathetic nervous hyperactivity has been suggested to decrease aerobic capacity of skeletal muscles based on reduced capillarisation[8] and reduced red blood cell flux[9] leading to a shift in muscle fibre type towards a lower content on type I fibres.[10] The ensuing anaerobic muscle metabolism leads to increased muscle fatiguability[11] and acidosis already at low levels of exercise, which trigger exaggerated responses in ventilation.[12] Hyperventilation, on the other hand, is well known to stimulate sympathetic nervous activity, and so the vicious circle of sympathetic nervous activity driving hyperventilation and hyperventilation activating sympathetic nervous activity continues.[13] This suggests that hyperventilation may not only be a consequence of poor left ventricular (LV) function, but also a driver.

Besides pharmaceutical therapies and electrophysiological interventions, exercise therapy has been found to have beneficial effects on hemodynamic and ventilatory parameters in HFrEF[14] and HFpEF patients alike.[15] The main mechanisms of exercise are thought to be reduced peripheral resistance and hence cardiac afterload by improvement of endothelial function, increased capillarisation leading to improved oxygenation of skeletal muscles and improved aerobic metabolism.[16] Despite the beneficial effects of exercise training in both, centre-based and home-based settings,[17, 18] adherence to physical activity has been found to be poor amongst HFrEF patients.[19] Surprisingly, few studies have targeted ventilation directly with therapeutic approaches. Only three studies have assessed the effects of slow-breathing training on cardiorespiratory function.[20, 21] These studies found improved physical function, reduced blood and pulmonary arterial pressure, increased ejection fraction (EF),[20, 22] improved ventilatory efficiency[20] and reduced sleep apnoea.[22] Further, they found improved regulation of the autonomic nervous system by reducing sympathetic drive and increasing vagal activity.[23] It is unknown whether slow breathing may increase PaCO2 sufficiently to change the sensitivity or set point of chemoreceptors. On the other hand, apnoea training has been found to lead to large changes in PaCO2 levels tolerated by chemoreceptors at rest and during exercise.[24, 25] However, to date there are no published studies that have implemented apnoea into a breathing training in HF patients. Further, previous studies have not investigated whether the effect of slow breathing on improving the V̇E/V̇CO2 slope was due to a chronic increase in PaCO2 or a decrease in ventilatory dead space.

HYPOTHESIS

The investigators hypothesise that a 12-week training with nasal slow breathing followed by end-expiratory apnoea based on education, centre-based introduction and home-based 15 min/day breathing training will be effective at reducing the exaggerated ventilatory response to exercise.

METHODS

Study design

Prospective randomised controlled study. Eligible patients are identified during their yearly check-up at the Heart Failure Clinic and Preventive Cardiology of the Inselspital in Bern. Patients will be randomised 1:1 (stratified for HFrEF/HFpEF and sex) to an intervention and control group. Patients in the intervention group perform the breathing training additionally to standard care and those in the control group receive standard care and are offered the breathing training after the end of the study. The study design and breathing intervention have been developed with direct input by a patient group (from pilot study).

In an additional cross-sectional substudy, the same measurements of the RCT are performed in a group of 15 patients after acute or chronic coronary syndrome (ACS/CCS) with inefficient ventilation, 15 healthy age-matched and 15 healthy young controls. Further, the cross-sectional substudy compares pulmonary gas exchange and breathing patterns during 5 min of oral versus 5 min of nasal breathing during submaximal continuous exercise in the HF, ACS/CCS, old healthy, and young healthy groups.

Breathing intervention

The respiratory pattern modulation training is performed at home for 12 weeks twice daily for 15 min per session and consists of three components: 1) education on abnormal ventilation in heart failure, the effect of ventilation on PaCO2 and the autonomous nervous system, and chemoreceptor sensitivity; 2) 1-3 sessions of guided and monitored face-to-face training with slow nasal abdominal breathing and intermittent apnoea supported by the Healer vest (L.I.F.E., Milan, Italy) measuring electrocardiogram (ECG), and chest excursions at the level of the xiphoid, thoracic manubrium, and abdomen; 3) independent home-based apnoea training supported by hand-outs, videos and weekly phone calls to monitor progress and adherence, answer questions and encourage further progression with duration of breath-hold.

Measurements

Measurements are performed during visit 1 before and visit 2 at the end of the intervention period.

Cardiopulmonary exercise testing (CPET)

CPETs are performed on a cycle ergometer according to the recommendations of the American Heart Association.[38] Ramp tests are performed as previously described.[31] O2 consumption and CO2 production will be measured continuously in an open spirometric system (Quark, Cosmed, Rome, Italy) and registered as average values over 8 breaths. Every 2 min, patients are asked about their perception of dyspnoea on the modified Borg scale. V̇E/V̇CO2 slope from rest to ventilatory threshold 2 (VT2), peak V̇O2 and V̇O2 at VT1 are determined as previously described.[31]

Blood analyses

Blood samples are obtained from the antecubital vein for analysis of haemoglobin and NT-proBNP. Arterialized blood are extracted from the ear lobe at rest and peak exercise for analysis of PaCO2, oxygen (PaO2), bicarbonate and pH.

Sensitivity of chemoreceptors

The sensitivity of chemoreceptors is measured by a rebreathing protocol.[39] The subjects are resting supine and breathe through a mouthpiece of an open spirometric system (Innocor, Cosmed, Rome, Italy). With the 3-way-valve open to room air, the test begins with 2-5 min of hyperventilation, allowing end-tidal partial CO2 pressure (PETCO2) to drop. Following hyperventilation, the subject breathes comfortably, while the 3-way-valve is switched to the rebreathing bag. Equilibration of PCO2 in bag, lungs, and arterial blood to mixed venous blood is achieved by taking three deep breaths. During the following minutes, PETCO2 is allowed to rise, while PETO2 is clamped at 150 mmHg during hyperoxic testing, and at 50 mmHg during a second, hypoxic test run by feeding 100% O2 into the circuit by a port at the rebreathing bag. Central and peripheral chemoreflex responses to CO2 are estimated by the difference between hyperoxic and hypoxic ventilatory response.[40, 41]

Patient reported outcomes

The Kansas City Cardiomyopathy Questionnaire (KCCQ) are filled in during visit 1 and visit 2 to assess quality of life and dyspnoea. During visit 2, a structured interview is performed with the patient to assess feasibility and barriers with the breathing training. Adherence to training is monitored based on verbal information by the patients during the weekly phone calls.

Heart rate variability (HRV) and breathing frequency (BF)

HRV is measured from 24-hour ECG recorded with the Healer vest (L.I.F.E., Milan, Italy) and analysed from a segment during a deep sleep phase as previously described by the investigators' group.[42] Low-frequency power (LF, ms2, 0.04-0.15 Hz), high-frequency power (HF, ms2, 0.15-0.4 Hz), and the LF/HF are analysed [43]. BF is measured by strain gauges from Healer vest.

Submaximal tests of cross-sectional substudy

After a 15 min break following the CPET ramp test, patients cycle 5 min at 50% of peak power output as assessed during the ramp test with exclusively nasal, and 5 min with exclusively oral breathing in randomised order, with a 15 min break between the two tests. Pulmonary gas exchange parameters and breathing pattern are measured and compared between the two breathing modes and between the four groups (HF, ACS/CCS, old healthy, young healthy).

OUTCOMES

Primary outcome is V̇E/V̇CO2 slope analysed by ANCOVA with repeated measures corrected for baseline values and EF and sex.

Secondary outcomes are the nadir of the V̇E/V̇CO2 ratio, breathing pattern, VD/VT, peak V̇O2, V̇O2 at VT1, resting PETCO2, peripheral and central chemoreceptor sensitivity, arterial blood gases, NT-proBNP, heart rate, HRV, ventricular premature beats from 24-hour ECG, KCCQ, feasibility and adherence.

Outcomes of cross-sectional study are VE/VCO2 ratio, VE, VO2, BF, VT, PetCO2, PetO2, O2/HR and rapid shallow breathing index between nasal and oral breathing.

REFERENCES

1. Agostoni P, Guazzi M. Exercise ventilatory inefficiency in heart failure: some fresh news into the roadmap of heart failure with preserved ejection fraction phenotyping. European journal of heart failure 2017; 19(12): 1686-9.
2. Ponikowski P, Francis DP, Piepoli MF, et al. Enhanced ventilatory response to exercise in patients with chronic heart failure and preserved exercise tolerance: marker of abnormal cardiorespiratory reflex control and predictor of poor prognosis. Circulation 2001; 103(7): 967-72.
3. Myers J, Arena R, Oliveira RB, et al. The lowest VE/VCO2 ratio during exercise as a predictor of outcomes in patients with heart failure. Journal of cardiac failure 2009; 15(9): 756-62.
4. Nadruz W, Jr., West E, Sengelov M, et al. Prognostic Value of Cardiopulmonary Exercise Testing in Heart Failure With Reduced, Midrange, and Preserved Ejection Fraction. Journal of the American Heart Association 2017; 6(11).
5. Johnson RL, Jr. Gas exchange efficiency in congestive heart failure. Circulation 2000; 101(24): 2774-6.
6. Chua TP, Clark AL, Amadi AA, et al. Relation between chemosensitivity and the ventilatory response to exercise in chronic heart failure. Journal of the American College of Cardiology 1996; 27(3): 650-7.
7. Scott AC, Davies LC, Coats AJ, et al. Relationship of skeletal muscle metaboreceptors in the upper and lower limbs with the respiratory control in patients with heart failure. Clinical science (London, England : 1979) 2002; 102(1): 23-30.
8. Duscha BD, Kraus WE, Keteyian SJ, et al. Capillary density of skeletal muscle: a contributing mechanism for exercise intolerance in class II-III chronic heart failure independent of other peripheral alterations. Journal of the American College of Cardiology 1999; 33(7): 1956-63.
9. Hirai DM, Musch TI, Poole DC. Exercise training in chronic heart failure: improving skeletal muscle O2 transport and utilization. Am J Physiol Heart Circ Physiol 2015; 309(9): H1419-39.
10. Sullivan MJ, Duscha BD, Klitgaard H, et al. Altered expression of myosin heavy chain in human skeletal muscle in chronic heart failure. Med Sci Sports Exerc 1997; 29(7): 860-6.
11. Schulze PC, Linke A, Schoene N, et al. Functional and morphological skeletal muscle abnormalities correlate with reduced electromyographic activity in chronic heart failure. Eur J Cardiovasc Prev Rehabil 2004; 11(2): 155-61.
12. Piepoli M, Clark AL, Volterrani M, et al. Contribution of muscle afferents to the hemodynamic, autonomic, and ventilatory responses to exercise in patients with chronic heart failure: effects of physical training. Circulation 1996; 93(5): 940-52.
13. Coats AJ, Clark AL, Piepoli M, et al. Symptoms and quality of life in heart failure: the muscle hypothesis. Br Heart J 1994; 72(2 Suppl): S36-9.
14. Tucker WJ, Lijauco CC, Hearon CM, Jr., et al. Mechanisms of the Improvement in Peak VO(2) With Exercise Training in Heart Failure With Reduced or Preserved Ejection Fraction. Heart Lung Circ 2018; 27(1): 9-21.
15. Fu TC, Yang NI, Wang CH, et al. Aerobic Interval Training Elicits Different Hemodynamic Adaptations Between Heart Failure Patients with Preserved and Reduced Ejection Fraction. Am J Phys Med Rehabil 2016; 95(1): 15-27.
16. Hambrecht R, Niebauer J, Fiehn E, et al. Physical training in patients with stable chronic heart failure: effects on cardiorespiratory fitness and ultrastructural abnormalities of leg muscles. Journal of the American College of Cardiology 1995; 25(6): 1239-49.
17. Ruku DM, Tran Thi TH, Chen HM. Effect of center-based or home-based resistance training on muscle strength and VO(2) peak in patients with HFrEF: A systematic review and meta-analysis. Enferm Clin (Engl Ed) 2021.
18. Long L, Mordi IR, Bridges C, et al. Exercise-based cardiac rehabilitation for adults with heart failure. Cochrane Database Syst Rev 2019; 1(1): Cd003331.
19. Cooper LB, Mentz RJ, Sun JL, et al. Psychosocial Factors, Exercise Adherence, and Outcomes in Heart Failure Patients: Insights From Heart Failure: A Controlled Trial Investigating Outcomes of Exercise Training (HF-ACTION). Circulation Heart failure 2015; 8(6): 1044-51.
20. Parati G, Malfatto G, Boarin S, et al. Device-guided paced breathing in the home setting: effects on exercise capacity, pulmonary and ventricular function in patients with chronic heart failure: a pilot study. Circulation Heart failure 2008; 1(3): 178-83.
21. Lachowska K, Bellwon J, Narkiewicz K, et al. Long-term effects of device-guided slow breathing in stable heart failure patients with reduced ejection fraction. Clinical research in cardiology : official journal of the German Cardiac Society 2019; 108(1): 48-60.
22. Kawecka-Jaszcz K, Bilo G, Drożdż T, et al. Effects of device-guided slow breathing training on exercise capacity, cardiac function, and respiratory patterns during sleep in male and female patients with chronic heart failure. Pol Arch Intern Med 2017; 127(1): 8-15.
23. Lachowska K, Bellwon J, Moryś J, et al. Slow breathing improves cardiovascular reactivity to mental stress and health-related quality of life in heart failure patients with reduced ejection fraction. Cardiology journal 2020; 27(6): 772-9.
24. Roecker K, Metzger J, Scholz T, et al. Modified ventilatory response characteristics to exercise in breath-hold divers. International journal of sports physiology and performance 2014; 9(5): 757-65.

31. Marcin T, Trachsel LD, Dysli M, et al. Effect of self-tailored high-intensity interval training versus moderate-intensity continuous exercise on cardiorespiratory fitness after myocardial infarction: A randomized controlled trial. Ann Phys Rehabil Med 2021: 101490.

38. Fletcher GF, Ades PA, Kligfield P, et al. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation 2013; 128(8): 873-934.

39. Duffin J. Measuring the respiratory chemoreflexes in humans. Respir Physiol Neurobiol 2011; 177(2): 71-9.

40. Duffin J, Mohan RM, Vasiliou P, et al. A model of the chemoreflex control of breathing in humans: model parameters measurement. Respir Physiol 2000; 120(1): 13-26.

41. Guyenet PG. Regulation of breathing and autonomic outflows by chemoreceptors. Compr Physiol 2014; 4(4): 1511-62.

42. Herzig D, Eser P, Omlin X, et al. Reproducibility of Heart Rate Variability Is Parameter and Sleep Stage Dependent. Frontiers in physiology 2017; 8: 1100.

43. Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. European heart journal 1996; 17(3): 354-81.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association (NYHA) functional classes II and III
* LVEF either <50% or ≥50%
* V̇E/V̇CO2 slope ≥36, and/or a pattern of exercise oscillatory ventilation defined by established criteria
* Optimal guideline-directed medical therapy for >3 months
* Written informed consent

Exclusion Criteria:

* Heart failure decompensation within the preceding 3 months
* Non-cardiac conditions and comorbidities associated with hyperventilation like pulmonary diseases
* Inability or unwillingness to perform apnoea training

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Ventilation to carbon dioxide production slope | Change from before to after 12-week breathing intervention
  Ventilation to carbon dioxide production (VE/VCO2) slope during ramp test

SECONDARY OUTCOMES:
Nadir of ventilation to carbon dioxide production ratio | Change from before to after 12-week breathing intervention
  Nadir of ventilation to carbon dioxide production ratio during ramp test
Breathing frequency | Change from before to after 12-week breathing intervention
  Breathing frequency at rest
Pulmonary efficiency | Change from before to after 12-week breathing intervention
  Pulmonary deadspace ventilation to tidal ventilation (VD/VT)
Aerobic capacity | Change from before to after 12-week breathing intervention
  Oxygen consumption at the 1st ventilatory threshold during ramp test
Resting end-tidal carbon dioxide | Change from before to after 12-week breathing intervention
  Resting end-tidal carbon dioxide during resting spirometry
Chemosensitivity | Change from before to after 12-week breathing intervention
  Sensitivity (gain and threshold) of peripheral and central chemoreceptors to carbon dioxide during hypo- and hyperoxia
Arterialised blood bicarbonate | Change from before to after 12-week breathing intervention
  Bicarbonate of arterialised blood from the earlobe
Arterialised blood CO2 | Change from before to after 12-week breathing intervention
  CO2 of arterialised blood from the earlobe
Arterialised blood O2 | Change from before to after 12-week breathing intervention
  O2 of arterialised blood from the earlobe
Arterialised blood pH | Change from before to after 12-week breathing intervention
  PH of arterialised blood from the earlobe
Myocardial stress marker | Change from before to after 12-week breathing intervention
  NT-proBNP from venous blood as marker of myocardial stress
Heart rate variability | Change from before to after 12-week breathing intervention
  Heart variability at rest
Arrhythmia | Change from before to after 12-week breathing intervention
  Ventricular premature beats measured by 24-h electrocardiogram
Patient reported outcome | Change from before to after 12-week breathing intervention
  Kansas City Cardiomyopathy Questionnaire
Feasibility of breathing training | Change from before to after 12-week breathing intervention
  Feasibility of breathing training by patient interviews
Adherence | Change from before to after 12-week breathing intervention
  Adherence to breathing training by patient interviews

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Wilhelm, Prof. MD, Principal Investigator — Preventive Cardiology & Sports Medicine, Dept. of Cardiology, University Hospital Berne
Locations (1):
- Preventive Cardiology and Sports Medicine, Bern University Hospital, Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eser P, Kaesermann D, Calamai P, Kalberer A, Stutz L, Huber S, Duffin J, Wilhelm M. Excess ventilation and chemosensitivity in patients with inefficient ventilation and chronic coronary syndrome or heart failure: a case-control study. Front Physiol. 2025 Jan 22;15:1509421. doi: 10.3389/fphys.2024.1509421. eCollection 2024. PMID 39911179